CLINICAL TRIAL: NCT04833764
Title: Mechanisms of Deep Vein Thrombosis (DVT) and Vein Wall Fibrosis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Khanh Nguyen (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Khanh Nguyen, Assistant Professor, Portland VA Medical Center
Organization: Portland VA Medical Center (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: eIRB19051/M4069
Record Dates: First submitted 2021-04-02; First posted 2021-04-06 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Post-thrombotic Syndrome; Deep Vein Thrombosis Leg
Keywords: Contact pathway inhibition; Coagulation factor XI inhibition; Anticoagulant; Deep vein thrombosis; Venous thrombosis
MeSH Terms: conditions — Postthrombotic Syndrome; Venous Thrombosis | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: This is a prospective, single arm Phase 1/Phase 2 study of patients with lower extremity DVT. Phase 1 will assess safety and tolerability of xisomab 3G3 in patients with lower extremity DVT on standard rivaroxaban therapy in 12-18 subjects. Three doses of xisomab 3G3 (42, 126, or 252 mg IV) will be tested to determine the maximum tolerated dose (MTD) with the dose limiting toxicity as any major bleeding or serious adverse event. Phase 2 will assess the efficacy of xisomab 3G3 for the prevention of PTS and compare the 1 year incidence of PTS as determined by the Villalta score in patients with lower extremity DVT on standard rivaroxaban therapy in 30 study participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rosuvastatin (Experimental): Subjects will receive 20 mg daily dose of rosuvastatin for at least 3 months
  Interventions: Drug: Rosuvastatin

INTERVENTIONS:
Drug: Rosuvastatin — Oral administration of 20 mg rosuvastatin for at least 3 months

SUMMARY:
The goal of this study is to determine the safety and tolerability or efficacy of adjunctive treatments (including rosuvastatin 20 mg daily) in combination with standard anticoagulation therapy (Factor Xa inhibitors) in patients with lower extremity deep vein thrombosis (DVT). The efficacy of adjunctive treatments to prevent the development of post thrombotic syndrome (PTS) after DVT will be evaluated.

DETAILED DESCRIPTION:
Post-thrombotic syndrome (PTS) is a significant complication that occurs up to 75% of patients after DVT. Rosuvastatin is a HMGCoA reductase inhibitor that has anti-inflammatory effects. In this study, the investigators will evaluate the safety and tolerability of combination standard anticoagulation therapy (e.g. Factor Xa inhibitor, rivaroxaban, apixaban) and three months of 20 mg dose of rivaroxaban and its efficacy as prophylaxis against PTS after lower extremity DVT. After the diagnosis of lower extremity DVT with either duplex venous ultrasound or other imaging, study participants will initiate standard rivaroxaban therapy as per standard medical care. All consented participants in this trial will receive three months of rosuvastatin (20 mg daily dose). Assessment of post thrombotic syndrome follow up will continue for 365 days from the time of DVT diagnosis or until resolution or stabilization of any clinically significant drug related adverse event, after which they will be considered off-study.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Diagnosis of a first episode of acute proximal leg DVT within 4 weeks of initial DVT diagnosis and without symptomatic pulmonary embolism (PE)
* Must have ECOG performance status ≤ 2
* Expected life expectancy of >2 years
* Before initiation of anticoagulation, must have adequate platelet count: Platelet count > 100 x 10^9/L,
* Before initiation of anticoagulation, must have adequate hemoglobin (Hgb) count: Hgb > 9 mg/DL
* Before initiation of anticoagulation, must have normal INR and PTT: INR ≤ 1.5 and aPTT≤40

Exclusion Criteria:

* Concurrent participation in another therapeutic clinical trial
* History of prior DVT in the previous 2 years
* Recurrent deep vein thrombosis (DVT)
* Established post thrombotic syndrome (PTS)
* Limb-threatening circulatory compromise
* Pulmonary embolism with hemodynamic compromise
* Deranged baseline coagulation profile before initiation of anticoagulation: INR > 1.5 or aPTT prolonged >40
* Active bleeding within last 3 months
* Anemia with Hemoglobin<9 mg/dL
* Thrombocytopenia with platelets < 100,000/ml
* Previously documented hypersensitivity to either the drug or excipients
* Any contraindication to anticoagulation or allergy to factor V inhibitors or ferumoxytol
* Any contraindication to magnetic resonance imaging (MRI) including metal implants or claustrophobia
* Severe hepatic impairment as defined by Childs-Pugh Class B or C
* Severe renal impairment with CrCl<30 ml/min,
* Taking any P-GP or strong CYP3A4 inhibitors or inducers
* History of major bleeding including history of gastrointestinal bleeding or intracranial bleeding
* Known history of bleeding diathesis
* History of chronic atrial fibrillation or stroke
* History of active cancer or malignancy within 1 year,
* Life expectancy <2 years.
* Patients requiring emergent or urgent surgery or procedures within the first 3 months of the study that cannot be postponed will be excluded.
* Patients who are breastfeeding or anticipate pregnancy
* Participant is pregnant or breastfeeding
* Participant is a prisoner (protected population)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Post-thrombotic syndrome | 365 day
  Incidence of post-thrombotic syndrome as measured by the Villalta Scale (score = or > 4). Minimum score=0, Maximum score=33, and a higher score indicates worse outcome.

SECONDARY OUTCOMES:
Severity of post-thrombotic syndrome (PTS) | 365 day
  Villalta score severity of post-thrombotic syndrome

CONTACTS AND LOCATIONS:
Overall Officials: Khanh P Nguyen, MD, Principal Investigator — Portland VA Medical Center
Locations (1):
- VA Portland Health Care System (VAPORHCS), Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No